CLINICAL TRIAL: NCT05378399
Title: SmartSteps: A Context-Aware, Pre-Exposure Prophylaxis Adherence Intervention for Individuals With Substance Use Disorder
Brief Title: SmartSteps: A Context-Aware, PrEP Adherence Intervention for Individuals With Substance Use Disorder
Acronym: SmartSteps
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Gilead Sciences (Industry); The Fenway Institute (Other)
Responsible Party: Principal Investigator, Peter R Chai MD, Emergency Medicine Physician, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021P003683
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: HIV Infections; Substance Use; Adherence, Medication; Adherence, Treatment
Keywords: Pre-Exposure Prophylaxis; Substance Use; Digital Pill System; Adherence; HIV Prevention
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders; Medication Adherence; Treatment Adherence and Compliance | interventions — emtricitabine tenofovir alafenamide; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Digital Pills and Beiwe (Experimental): Participants will take one PrEP digital pill per day, for 60 days total, while using the ID-Cap digital pill system and Beiwe digital phenotyping app.
  Interventions: Drug: Descovy or Truvada; Device: ID-Cap System; Device: Beiwe

INTERVENTIONS:
Drug: Descovy or Truvada — Descovy or Truvada prescribed with digital pills for PrEP
Device: ID-Cap System — Digital pills overencapsulating Descovy or Truvada for PrEP
  Other Names: digital pill
Device: Beiwe — Digital phenotyping app

SUMMARY:
This is a single-arm, observational study of HIV-negative MSM with substance use disorder. Those who meet pre-screening criteria will attend a Screening Visit (Visit 1), where the informed consent process will be conducted and study eligibility will be confirmed. Eligible participants will attend three additional visits over the course of the study - the Enrollment Visit (Visit 2), Month 1 Visit (Visit 3), and Month 2 Visit (Visit 4). Participants will take one PrEP digital pill per day, for 60 days total, while using the digital pill system (DPS) and Beiwe, a digital phenotyping app. On nonadherent days, participants will receive brief surveys prompting them to report the reasons for their missed dose, as well as their engagement in substance use and sexual activity. Timeline followback will be conducted at the Month 1 and Month 2 Visits to understand the context of any nonadherence. Qualitative user experience exit interviews and dried blood spots (DBS) will be conducted at the Month 2 Visit.

DETAILED DESCRIPTION:
This study will develop a dataset of annotated smartphone usage in the context of PrEP adherence and nonadherence. In order to understand smartphone context, the investigators will utilize a digital pill system (DPS) to measure real-time PrEP ingestion events. Eligibility will be confirmed during the Screening Visit (Visit 1). During the Enrollment Visit (Visit 2), participants will complete a baseline quantitative assessment (e.g., sociodemographics, sexual history, attitudes about technology), receive training on the operation of the DPS and Beiwe, and will ingest their first digital pill dose under observation by study staff. Participants will be instructed to take one PrEP pill once daily while using the DPS and Beiwe app for 60 days. Participants will return for a study visit at the end of month one (Visit 3) for a refill of digital pills. Following a 24-hour period which no PrEP ingestion is detected by the DPS, participants will receive a brief online substance use and sexual risk survey, which will inform specific contexts of nonadherence. At the Month 1 Visit (Visit 3) and Month 2 Visit (Visit 4), timeline followback discussions will be conducted to better understand the context of any PrEP nonadherence events detected by the DPS, and phenotypic data collected by the Beiwe app, during the prior 30 days. At the Month 2 (Visit 4), the investigators will administer a blood draw for dried blood spot (DBS) testing to measure participants' PrEP adherence and compare it against adherence detected by the DPS. To gain insight into user experiences operating the DPS and Beiwe app as part of the study, the investigators will conduct the semi-structured qualitative exit interviews with participants at Month 2 (Visit 4).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Cisgender male
3. Has sex with men
4. HIV negative
5. On PrEP or initiating PrEP (including switching from 2-1-1 or "on-demand" PrEP dosing to once-daily dosing)
6. Moderate risk score on ASSIST substance use screener (11-26 for alcohol, 4-26 for all other substances) or higher
7. Qualifying laboratory testing for PrEP: Cr clearance in past 3 months, HBV vaccination, liver function tests
8. Owns a smartphone with Android or iOS

Exclusion Criteria:

1. Does not speak English
2. History of Crohn's disease or ulcerative colitis
3. History of gastric bypass or bowel stricture
4. History of GI malignancy or radiation to abdomen
5. Allergy to gelatin, silver, or zinc (components of digital pill)
6. Allergy to PrEP
7. Not willing to operate DPS or Beiwe app

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender men who have sex with men
Enrollment: 40 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
PrEP Adherence Patterns | After Month 2 Visit
  Percentage adherence to PrEP and adherence patterns over the course of 60 days, as detected by the ID-Cap digital pill system (DPS).
Correlation of PrEP Adherence with Digital Phenotyping Patterns | After Month 2 Visit
  Comparison of digital phenotyping data, as detected by Beiwe, on PrEP-adherent versus PrEP-nonadherent days, as detected by the digital pill system (DPS).

SECONDARY OUTCOMES:
Correlation of PrEP Adherence with DBS Concentrations | After Month 2 Visit
  Correlation of PrEP adherence patterns, as detected by the digital pill system (DPS), with tenofovir diphosphate concentrations in dried blood spots (DBS).
Acceptability of DPS and Digital Phenotyping App | After Month 2 Visit
  User acceptance of and willingness to interact with the digital pill system (DPS) and Beiwe digital phenotyping app, as assessed via qualitative exit interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Peter R Chai, MD MMS, Principal Investigator — Brigham and Women's Hopsital
Locations (1):
- Fenway Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No